CLINICAL TRIAL: NCT03926845
Title: Efficacy and Tolerability of an Isobutylamido-thiazolyl-resorcinol Cream 0.2% for Facial Hyperpigmentation, A Randomized Double-blind and Vehicle-Controlled Study
Brief Title: Efficacy and Tolerability of an Isobutylamido-thiazolyl-resorcinol Cream 0.2% for Facial Hyperpigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Dermatology, Thailand (Other Government)
Collaborators: Beiersdorf (Thailand) Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Chinmanat Lekhavat, Assistant Director, Institute of Dermatology, Thailand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 013/2562
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Facial Hyperpigmentation
Keywords: Isobutylamido-thiazolyl-resorcinol

STUDY DESIGN:
Intervention Model Description: This is a randomized, vehicle controlled, double-blind study and is performed at the Institute of Dermatology. Subjects are randomized into 2 groups by a computer prior to the start of the study - group 1 receives Isobutylamido-thiazolyl-resorcinol 0.2% cream and group 2 receives vehicle cream for 12 weeks. Both Study products have to be applied twice daily.Total of 4 clinical sessions are carried out in order to evaluate Isobutylamido-thiazolyl-resorcinol 0.2% efficacy and tolerability at week 4, 8 and 12. Subjects and investigators are blinded about allocation. The appearance of the vehicle formulation was similar to the verum formulation and could not be distinguished neither by patients nor by the investigator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isobutylamido-thiazolyl-resorcinol Cream 0.2% (Active Comparator): The cream contains 0.2% Isobutylamido-thiazolyl-resorcinol.
  Interventions: Other: Isobutylamido-thiazolyl-resorcinol Cream 0.2%
- Vehicle (Placebo Comparator): The cream contains no active ingredients.
  Interventions: Other: Vehicle

INTERVENTIONS:
Other: Isobutylamido-thiazolyl-resorcinol Cream 0.2% — Each bottle contains Isobutylamido-thiazolyl-resorcinol cream 0.2% to be applied on the entire face twice daily for 12 weeks.
  Arms: Isobutylamido-thiazolyl-resorcinol Cream 0.2%
Other: Vehicle — Each bottle contains vehicle cream to be applied on the entire face twice daily for 12 weeks.
  Arms: Vehicle

SUMMARY:
Facial hyperpigmentation is a common skin issue that can cause embarrassment and affect the quality of life in majority of people. The investigators are conducting a research to study an efficacy and tolerability of Isobutylamido-thiazolyl-resorcinol 0.2% in lightening of the facial hyperpigmentation in comparison to vehicle intervention in 4, 8 and 12-week period. The ultimate goal is to provide the best cosmetic cream to improve the quality of life of people who suffer from facial hyperpigmentation.

DETAILED DESCRIPTION:
Facial hyperpigmentation is a skin issue that occurs frequently in people with darker skin types. Studies show that the prevalence of facial hyperpigmentation is related to ethnicity and is accounted for up to 40%of the total population. The pathogenesis of facial hyperpigmentation is still unclear, but several factors seem to contribute such as ultraviolet radiation, female hormones, and genetics, which increase melanin production in the skin cells, specifically the epidermal melanocyte, and dermal melanophage. Hyperpigmentation can be embarrassing and affect the quality of life in the pertained individuals.

Tyrosinase enzyme plays a key element in melanin production which causes dark areas. In 2018, several studies have reported a new cosmetic product using Isobutylamido-thiazolyl-resorcinol (Beiersdorf AG, Hamburg, Germany) in facial hyperpigmentation. In vitro studies found that in melanocyte culture, Isobutylamido-thiazolyl-resorcinol inhibit melanin production. Studies discovered that Isobutylamido-thiazolyl-resorcinol 0.2% can reduce facial hyperpigmentation within 4 weeks. Hyperpigmentation begin to fade away within 12 weeks of daily application.

The objective is to study efficacy and tolerability of a cosmetic formulation with Isobutylamido-thiazolyl-resorcinol 0.2% compared to its vehicle in facial hyperpigmentation after 4, 8 and 12-week.

This is a randomized double-blind and vehicle-controlled study. Two hundred subjects both male and female 18 years or older with facial hyperpigmentation are recruited in the study. The study was performed at the Institute of Dermatology, Bangkok, Thailand. Subjects agree to attend monthly sessions every 4 weeks for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are Thai adults age 18 years old and above .
2. Subjects suffer from facial hyperpigmentation for at least 10 years, with or without freckles, lentigo or dark sports.
3. Subjects must be able to attend monthly sessions in the period of 12 weeks session.
4. Subjects must refrain from using other whitening cream such as hydroquinone, azelaic acid, kojic acid, arbutin, glycolic acid or any other creams which whiten the skin including chemical peel or whitening pills such as Tranexamic acid at least 1 month before the trial.
5. Subjects must refrain from receiving both ablative and nonablative laser treatment at least 3 months before the trial.
6. Subjects who can apply sun screen with UVA and UVB protection that has a minimum of SPF30 daily.

Exclusion Criteria:

1. Subjects who have conditions such as Lichen planus pigmentosus, Pigmented contact dermatitis, Photosensitivity, Ashy dermatosis, Dermal melanosis, e.g. Nevus of Hori, Nevus of Ota, Dermal melanocyte hamartoma
2. Subjects with a congenital disease which darkens skin tone, e.g. Addison's disease, Cushing's syndrome and Thyrotoxicosis
3. Subjects with a congenital or serious disease with unpredictable symptoms such as Cirrhosis, cardiovascular diseases, Neurological diseases, gastrointestinal disease, Reproductive system diseases, Cancer and Psychiatric diseases.
4. Subjects who take pills that might cause hyperpigmentation such as chemotherapy, Amiodarone, Chlorpromazine, Hydroxychloroquine, Gold, Birth control pills (if related to causing hyperpigmentation issue)
5. Female subjects with pregnancy and breastfeeding.
6. Subjects who are allergic to chemical compound in the cream such as Alcohol denat, Phenoxyethanol or fragrance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Color assessment of facial hyperpigmentation by Color Analysis program will be evaluated every visit. | 12 weeks
  Each visit, photos are taken on all patients by VISIA-CR system camera on 3 positions of the face, straight and 37* on both sides with standard unfiltered and cross polarized lens. Each time the photos are filed and the colors are analyzed in order to be compared the changes between visits.
Physician's Global Assessment of facial hyperpigmentation will be evaluated every visit. | 12 weeks
  Evaluate the changes of facial hyperpigmentation by global assessment score: 0=Completely clear,1=Almost clear, 2=Marked improved, 3=Moderate improved, 4=Slight improved, 5=No change, 6=Worse
Patient's Global Assessment of facial hyperpigmentation will be evaluated every visit. | 12 weeks
  Evaluate the changes of facial hyperpigmentation by global assessment score: 0=Completely clear,1=Almost clear, 2=Marked improved, 3=Moderate improved, 4=Slight improved, 5=No change, 6=Worse
Patient's Self-Grading of facial hyperpigmentation will be evaluated every visit. | 12 weeks
  Visual self-grading by patients from 1 to 10 by 1 is the least and 10 is the most in the criteria of evenness, spots and skin clarity
Evaluate side effects of Isobutylamido-thiazolyl-resorcinol cream 0.2% or vehicle cream every visit. | 12 weeks
  All patients are asked about the side effects of using the cream such as eczema, hypopigmentation, and redness.

CONTACTS AND LOCATIONS:
Overall Officials: Chinmanat Lekhavat, MD, Principal Investigator — Institute of Dermatology
Locations (1):
- Institute of Dermatology, Ratchathewi, Bangkok, Thailand

REFERENCES:
- [Background] Briganti S, Camera E, Picardo M. Chemical and instrumental approaches to treat hyperpigmentation. Pigment Cell Res. 2003 Apr;16(2):101-10. doi: 10.1034/j.1600-0749.2003.00029.x. PMID 12622786
- [Background] Rossi AM, Perez MI. Treatment of hyperpigmentation. Facial Plast Surg Clin North Am. 2011 May;19(2):313-24. doi: 10.1016/j.fsc.2011.05.010. PMID 21763992
- [Background] Ortonne JP, Pandya AG, Lui H, Hexsel D. Treatment of solar lentigines. J Am Acad Dermatol. 2006 May;54(5 Suppl 2):S262-71. doi: 10.1016/j.jaad.2005.12.043. PMID 16631967
- [Background] Mann T, Gerwat W, Batzer J, Eggers K, Scherner C, Wenck H, Stab F, Hearing VJ, Rohm KH, Kolbe L. Inhibition of Human Tyrosinase Requires Molecular Motifs Distinctively Different from Mushroom Tyrosinase. J Invest Dermatol. 2018 Jul;138(7):1601-1608. doi: 10.1016/j.jid.2018.01.019. Epub 2018 Feb 7. PMID 29427586
- [Background] Lacz NL, Vafaie J, Kihiczak NI, Schwartz RA. Postinflammatory hyperpigmentation: a common but troubling condition. Int J Dermatol. 2004 May;43(5):362-5. doi: 10.1111/j.1365-4632.2004.02267.x. No abstract available. PMID 15117368
- [Background] Espin JC, Varon R, Fenoll LG, Gilabert MA, Garcia-Ruiz PA, Tudela J, Garcia-Canovas F. Kinetic characterization of the substrate specificity and mechanism of mushroom tyrosinase. Eur J Biochem. 2000 Mar;267(5):1270-9. doi: 10.1046/j.1432-1327.2000.01013.x. PMID 10691963
- [Background] Weatherall IL, Coombs BD. Skin color measurements in terms of CIELAB color space values. J Invest Dermatol. 1992 Oct;99(4):468-73. doi: 10.1111/1523-1747.ep12616156. PMID 1402005
- [Derived] Lekhavat C, Rojanamatin J, Suphannaphong M, Kolbe L. Efficacy and Tolerability of 0.2% Thiamidol Cream for Facial Hyperpigmentation: A Randomized, Double-Blind, and Vehicle-Controlled Study. Dermatol Ther (Heidelb). 2026 Jan 21. doi: 10.1007/s13555-025-01649-y. Online ahead of print. PMID 41566113